CLINICAL TRIAL: NCT03068429
Title: Fear Conditioning, Extinction and Recall in Healthy Subjects and in Obsessive-compulsive Disorder Patients Pre and Post Treatment With Sertraline.
Brief Title: Fear Conditioned Response in Healthy Subjects and in OCD Patients Pre and Post Treatment With Sertraline.
Acronym: FEARCON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Juliana Belo Diniz, Psychiatrist, principal investigator, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0182/11
Record Dates: First submitted 2017-02-22; First posted 2017-03-01 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: obsessive-compulsive disorder; fear conditioning; functional neuroimaging; sertraline
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Sertraline

STUDY DESIGN:
Intervention Model Description: 4-weeks open label trial of sertraline up to 200mg/day treatment for obsessive compulsive disorder
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sertraline open label (Experimental): Sertraline hydrochloride up to 200mg/day or maximum tolerated dosage for 4-weeks.
  Interventions: Drug: Sertraline Hydrochloride

INTERVENTIONS:
Drug: Sertraline Hydrochloride — first week: sertraline hydrochloride 50mg/day, second week: sertraline hydrochloride 100mg/day, third week: sertraline hydrochloride 150mg/day, fourth week: sertraline hydrochloride 200mg/day OBS.: Other SSRIs (fluoxetine, paroxetine, escitalopram) with equivalent dosage schedules can be used if patients report prior intolerance to sertraline
  Other Names: sertraline 50mg; zoloft

SUMMARY:
24 OCD patients and 24 healthy subjects will be submitted to a two-day fear conditioning paradigm during acquisition of functional magnetic resonance imaging (fMRI). OCD patients will be submitted to the paradigm at two timepoints: baseline and 4 weeks after treatment initiation with sertraline up to 200mg/day or maximum tolerated dosage. OCD patients are expected to demonstrate worsened extinction retention compared to healthy subjects at baseline. Sertraline treatment is expected to improve extinction retention compared to baseline and to normalize the brain regions being recruited with the conditioned stimuli presented during the recall phase.

DETAILED DESCRIPTION:
Fear conditioning paradigms are used to investigate the learning process of the fear response in patients with psychiatric disorders and healthy subjects. Patients with post traumatic stress disorder have been shown to fail to retrieve the memory of fear extinction during the recall phase of the fear conditioning paradigm when compared to healthy subjects. In one previous trial, obsessive-compulsive disorder (OCD) patients have demonstrated the same failure to recall extinction and the results from functional magnetic resonance imaging (fMRI) activation maps have shown different regions being recruited during recall when compared with healthy subjects. However, in that previous trial, some of the OCD patients included were already taking medication for OCD. In the current trial, we will evaluate 24 unmedicated OCD patients with a two-day fear conditioning paradigm before and after 4-weeks of treatment initiation with sertraline up to 200mg/day or maximum tolerated dosage. Sertraline is a first-line treatment option for OCD. At baseline, OCD patients will be compared to 24 healthy subjects. At post treatment, fear conditioning and fMRI results wil be compared to baseline. OCD patients are expected to demonstrate worsened extinction retention compared to healthy subjects at baseline. Sertraline treatment is expected to improve extinction retention compared to baseline and to normalize the brain regions being recruited with the conditioned stimuli presented during the recall phase. By "normalize" we mean that after treatment the regions being recruited will be the same as the ones recruited by healthy subjects during baseline, in other words, differences found at baseline regarding brain activation by the conditioned stimuli are expected to disappear after treatment.

Abbreviations: CS= conditioned stimuli, CS+= conditioned stimuli to shock, CS-=neutral conditioned stimuli, CS+E= extinguished conditioned stimuli to shock, CS+U=unextinguished conditioned stimuli to shock

ELIGIBILITY:
Inclusion Criteria:

Healthy controls

-willingness to participate in research

OCD patients

* willingness to participate in research
* main diagnosis of OCD (psychiatric clinical evaluation)
* minimum YBOCS (Yale Brown Obsessive-compulsive severity scale) score of 16 points

Exclusion Criteria:

Healthy controls

* any current psychiatric diagnosis according to evaluation using semi structured interview for DSM IV diagnoses (SCID I)
* any past psychiatric diagnoses except single major depression episode and simple phobia (evaluation by semi structure interview-SCID I)
* current use of psychotropic medications (last use has to be at least 3 months prior to study initiation)
* chronic use of any medications except vitamins and contraceptives
* MRI exclusionary criteria (metal implants, recently made tatoos, claustrophobia, etc)
* being pregnant

OCD patients

* comorbidity with neurodevelopmental disorders (autism, mental retardation), current psychotic disorders, current substance dependence or abuse, bipolar mood disorder according to evaluation using semi structured interview for DSM IV diagnoses (SCID I)
* current use of psychotropic medications (last use has to be at least 3 months prior to study initiation)
* MRI exclusion criteria(metal implants, recently made tatoos, claustrophobia, etc)
* being pregnant or at risk of becoming pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Main behavioral measure (extinction retention index) | Baseline for both groups (OCD and helthy subjects), change from baseline to 4 weeks after treatment initiation only for intervention group
  Equation: 100-((MEAN(2 first CS+E during recall)/MAXIMUM(2 last CS+E during extinction))*100)
Main functional neuroimaging measure | Baseline for both groups (OCD and helthy subjects), change from baseline to 4 weeks after treatment initiation only for intervention group
  ventro medial prefrontal cortex (vmPFC) activation during recall phase
Main treatment outcome measure | Change from baseline to 4 weeks after treatment initiation (only interventional group)
  Yale Brown Obsessive Compulsive Scale reduction (final score minus initial score)

SECONDARY OUTCOMES:
Main behavioral measure baseline comparison (extinction retention index OCD patients versus healthy subjects) | Baseline
  Equation: 100-((MEAN(2 first CS+E during recall)/MAXIMUM(2 last CS+E during extinction))*100)
Main functional neuroimaging measure (activation maps for contrast CS+E versus CS-during recall phase,OCD patients versus healthy subjects) | Baseline (all subjects)
  ventro medial prefrontal cortex (vmPFC) activation during recall phase
Secondary behavioral measure (learning- conditioning index, OCD patients pre and post treatment) | Change from baseline to 4 weeks after treatment initiation (only interventional group)
  Equation: MEAN(all CS+ during conditioning)-MEAN(all CS- during conditioning)
Secondary behavioral measure (learning- conditioning index, OCD patients versus healthy subjects) | Baseline (all subjects)
  Equation: MEAN(all CS+ during conditioning)-MEAN(all CS- during conditioning)
Secondary Behavioral Measure (context discrimination index based on skin conductance, OCD patients pre and post treatment) | Change from baseline to 4 weeks after treatment initiation (only interventional group)
  Equation: MEAN(first two CS+U during renewal)-MEAN(first two CS+U during recall)
Secondary Behavioral Measure (context discrimination index based on skin conductance, OCD patients versus healthy subjects) | Baseline (all subjects)
  Equation: MEAN(first two CS+U during renewal)-MEAN(first two CS+U during recall)
Secondary functional neuroimaging measure (functional activation maps for contrast CS+/CS- during conditioning phase, OCD patients pre and post treatment) | Change from baseline to 4 weeks after treatment initiation (only interventional group)
  Gain in amygdala activation during conditioning for CS+ presentations
Secondary functional neuroimaging measure (functional activation maps for contrast CS+/CS- during conditioning phase, OCD patients versus healthy subjects) | Baseline (all subjects)
  Gain in amygdala activation during conditioning for CS+ presentations
Secondary functional neuroimaging measure (functional activation maps for contrast CS+E/CS- during recall phase of baseline measurement, OCD patients versus healthy subjects) | Baseline (all subjects)
  Alternative activations (OCD patients versus controls), regions other than the vmPFC, activated with CS+ presentations during recall
Secondary functional neuroimaging measure (functional activation maps for contrast CS+E/CS- during recall phase comparing change between post and pre treatment) | Change between baseline and 4 weeks after treatment initiation (only interventional group)
  Alternative activations (OCD patients post treatment compared with baseline), regions other than the vmPFC, activated with CS+E presentations during recall

CONTACTS AND LOCATIONS:
Overall Officials: Juliana B Diniz, MD, PhD, Principal Investigator — Researcher
Locations (1):
- Institute of Psychiatry, Hospital das Clínicas, Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The spreadsheet with main results will be made available along main publication
Supporting Information: SAP, Analytic Code
Time Frame: Data is estimated to be available at study completion. Completion date is estimated to be july/2020.
Access Criteria: There will be no restrictions to acess of unindentified data results.